CLINICAL TRIAL: NCT07167836
Title: Effect of an Automated Clinical Pathway Utilizing Tailored Risk Stratification on Rates of Overdue Follow up and Outcomes in Patients With Inflammatory Bowel Disease
Brief Title: Automated Clinical Pathway for Inflammatory Bowel Disease Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Fudman, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: STU-2024-1013
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Disease; Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care pathway arm (Experimental): Use of an electronic medical record-based, risk-stratified tool that automates the identification of patients who are overdue for follow up and facilitates a proactive scheduling plan
  Interventions: Other: Electronic medical record-based care pathway
- Usual care (No Intervention): Standard disease management, monitoring, and follow-up as directed by clinical team

INTERVENTIONS:
Other: Electronic medical record-based care pathway — Participants will undergo initial automated risk stratification to direct tailored follow-up intervals. If exceeding the maximum time interval, participants in the intervention arm will be contacted by scheduling personnel using a standardized protocol to schedule a follow-up visit. In contrast, patients in the control arm who are overdue will not be made known to any staff and will not be proactively contacted, instead continuing to be managed according to standard of care. To maximize generalizability and understanding among staff and patients, risk stratification will be based on inflammatory bowel disease medication use.
  Arms: Care pathway arm

SUMMARY:
Pragmatic randomized controlled trial to evaluate the effect of an electronic medical record-based tool on improving on-time follow up and its effects on inflammatory bowel disease outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Alive patients with 2 or more visits to the UT Southwestern adult digestive disease clinic within 3 years of the date of trial commencement including at least one visit within 2 years, and
2. An active inflammatory bowel disease-specific medication, and
3. At least one of the following:

   1. Inflammatory bowel disease on the active problem list
   2. An inflammatory bowel disease invoice diagnosis at least twice in the 3 years prior to trial commencement
   3. An inflammatory bowel disease encounter diagnosis at least twice in the 3 years prior to trial commencement

Exclusion Criteria:

Patients not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of days overdue for completion of clinical follow up | 12 months
  Calculated on a per-patient basis with a denominator of 365 (days in the study period) and a numerator of days overdue for follow up. Definition of overdue follows a patient's risk stratification

SECONDARY OUTCOMES:
Composite clinical outcome: acute care utilization, steroid use, or inflammatory bowel disease-related surgery | 12 months
  Proportion of patients experiencing any event in the composite outcome of: a) acute care utilization, defined as combined incidence of visits to emergency rooms or admissions to the hospital; b) steroid use: incidence of new steroid prescriptions; and c) inflammatory bowel disease-related surgery
Proportion of patients with bowel-specific inflammatory assessment | 12 months
  The proportion of patients who completed a bowel-specific inflammatory assessment, defined as calprotectin, computed tomography or magnetic resonance enterography, or lower endoscopy (colonoscopy, sigmoidoscopy, pouchoscopy, ileoscopy)

OTHER OUTCOMES:
Proportion of patients with C-reactive protein measurement | 12 months
  Proportion of patients completing a measurement of C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No